CLINICAL TRIAL: NCT05152875
Title: Relationship Between Fungal Colonization and Severe Bronchopulmonary Dysplasia: Myth or Reality? Retrospective Study of Premature Infants Inferior to 29 Weeks of Gestation
Brief Title: Relationship Between Fungal Colonization and Severe Bronchopulmonary Dysplasia
Acronym: FunDyP
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/0060
Record Dates: First submitted 2021-11-19; First posted 2021-12-10 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2022-09

CONDITIONS: Bronchopulmonary Dysplasia; Extreme Prematurity; Fungal Infection
Keywords: Extremely premature infants; Bronchopulmonary dysplasia; fungal infection
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Mycoses | interventions — Biological Products

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: biological — fungal colonization by weekly cultures

SUMMARY:
The aim of this study is to determine if fungal colonization is associated to severe bronchopulmonary dysplasia in premature infants less than 29 weeks of gestation, and to determine if an association exists between fungal colonization and complications of prematurity and death.

DETAILED DESCRIPTION:
Fungal colonization is common in premature infants. Certain neonatal departments, routinely screen for fungal colonization by weekly cultures, while other departments perform fungal cultures solely in the presence of suggestive clinical or biological signs such as hyperleucocytosis, maternal vaginal candidiasis, sepsis and characteristic skin lesions. This neonatal colonization can progress to an invasive fungal infection leading to death and comorbidities. A relationship between fungal colonization and severe bronchopulmonary dysplasia is suspected.

ELIGIBILITY:
Inclusion Criteria:

* Premature infants inferior to 29 weeks of gestation screened for fungal colonization,
* Admitted in the neonatal department of Centre Hospitalier Sud Francilien,
* Between January 1st 2018 and December 31st 2020,
* Holders of parental authority informed of the study that are unopposed

Exclusion Criteria:

* Premature infants over 29 weeks of gestation, or term infants,
* Premature infants less than 29 weeks of gestation not screened for fungal colonization during their hospitalization,
* Premature infants with significant congenital malformations or genetic abnormalities,
* Premature infants inferior to 29 weeks of gestation deceased in delivery room.

Ages: 1 Day to 29 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Cohort will be selected among all extremely premature infants admitted between January 2018 and December 2020 in the neonatal intensive care unit of Centre Hospitalier Sud Francilien (Corbeil Essonnes 91, France)
Sampling Method: Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Severe bronchopulmonary dysplasia in premature infants inferior to 29 weeks of gestation | at 36 weeks corrected age
  Need of nCPAP, NIPPV, or nasal cannula ≥3 L/min with more than 30% of fraction inspired in Oxygen.

SECONDARY OUTCOMES:
Necrotizing enterocolitis | Day 0
  Necrotizing enterocolitis
Intraventricular haemorrhage grade 3 or 44 | Day 0
  Intraventricular haemorrhage grade 3 or 44
Retinopathy of prematurity | Day 0
  Retinopathy of prematurity
Invasive fungal infection | Day 0
  Invasive fungal infection
Death | Day 0
  Death

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Taher LAMOUCHI, MD, Principal Investigator — Centre Hospitalier Sud Francilien
Locations (1):
- LAMOUCHI Mohamed Taher, Corbeil-Essonnes, France, France

IPD SHARING:
Plan to Share IPD: No